CLINICAL TRIAL: NCT03600389
Title: Patient Priorities Care for Older Adults With Multiple Chronic Conditions Achieved Through Primary and Specialty Care Alignment: Patient Priorities Care (PPC)
Brief Title: Patient Priorities Care (PPC)
Acronym: PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The John A. Hartford Foundation (Other); Gordon and Betty Moore Foundation (Other); Robert Wood Johnson Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1601017608
Record Dates: First submitted 2018-05-01; First posted 2018-07-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Multiple Chronic Conditions
Keywords: Patient Health Priorities; Health Outcome Goals; Healthcare Preferences
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Interviewer and chart abstractor is blinded to the nature of the intervention and to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Implementing Patient Priorities Care) (Experimental): Aligning healthcare recommendations to achieve patients' specific health outcome goals within the context of what patients are willing and able to do.
  Interventions: Behavioral: Patient Priorities Care
- Control Arm (Not Implementing Patient Priorities Care) (No Intervention): Routine Care

INTERVENTIONS:
Behavioral: Patient Priorities Care
  Arms: Intervention Arm (Implementing Patient Priorities Care)

SUMMARY:
Patient Priorities Care aligns healthcare decision-making and care by all clinicians with patients' own health priorities. Patient Priorities Care involves not only the health outcome goals that patients want to achieve, but also their preferences for healthcare. This approach is about aligning what outcomes patients want from their healthcare with what they are willing and able to do to achieve these outcomes. The approach begins with a member of the healthcare team helping patients identify their health outcome goals and their care preferences and preparing them to interact with their clinicians around these goals and preferences. The goals and preferences are transmitted to the patient's clinicians who use them in decision-making and communication with the patient and other clinicians.

DETAILED DESCRIPTION:
Many older adults with Multiple Chronic Conditions receive conflicting recommendations and care that may be fragmented across clinicians. Older adults vary in what's most important when faced with tradeoffs and vary in the health-related activities they are willing and able to complete to achieve their desired outcomes. A potential solution to these problems is to move from decision-making predicated solely on disease-guidelines to decision-making based on achieving each patient's own specific health outcome goals (e.g., relief of symptoms sufficient to allow specific functional activity) within the context of what they are willing and able to do (i.e. care preferences) to achieve these outcomes.

The primary aims of the Patient Priorities Care (PPC) pilot is to assess the feasibility of aligning primary and specialty care to focus on the health priorities (i.e. specific and actionable outcome goals and care preferences) of older adults with multiple chronic conditions (MCC)

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Member of Pro-Health Practice for >=3 years
* Determined to be an appropriate candidate evidenced by ANY of the following:

  * Multiple Chronic Conditions (presence of >3 active health problems)
  * >10 medications
  * ≥ 1 hospitalization over the past year
  * ≥ 2 emergency department visits over the past year
  * Seen by >2 specialists (excluding GYN and eye) over the past year

Exclusion Criteria:

* End stage renal disease
* Unable to consent (e.g. dementia)
* In hospice or meeting hospice criteria
* Nursing home resident
* Not English speaking

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 414 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment Burden Questionnaire (TBQ) | 6-12 Months
  Measure to assess treatment burden among patients with one or more chronic conditions. Summary score is 0-150 with lower numbers indicating less burden. This is an exploratory study and the investigators will compare the intervention to control group to determine if the intervention group scores are lower on the TBQ (i.e. less burden).
Older Patient Assessment of Care for Chronic Conditions (O-PACIC) | 6-12 Months
  Measure to assess chronically-ill patients' perceptions of the degree to which health care delivery is integrated and coordinated. Summary score is 1-5 with higher score indicated greater integration. This is an exploratory study and the investigators will compare the intervention to control group to determine if the intervention group scores higher on O-PACIC (i.e. greater integration).
CollaboRATE | 6-12 Months
  Measure of shared decision making in clinical encounters. Summary score is 0-100 with higher score indicated greater shared decision making. This is an exploratory study and the investigator will compare the intervention to control group to determine if the intervention group scores higher on CollaboRATE (i.e. greater shared decision-making).
Health Care Utilization | 6-12 months
  Measures of changes in health care utilization drawn from review of patient medical records

SECONDARY OUTCOMES:
Older Patient Assessment of Care for Chronic Conditions (O-PACIC) subscales | 6-12 Months
  Sub-scales within the O-PACIC including patient activation (sub-scores range from 1-5 with higher score indicating greater activation), delivery system design/support (sub-scale score ranges from 1-5 with higher scores indicating greater system design/support), goal setting (sub-scale scores range from 1-5 with higher scores indicating improved goal setting), problem-solving/contextual counseling (sub-scale scores range from 1-5 with higher scores indicating improved problem-solving/contextual counseling), and follow-up/coordination (sub-scale scores range from 1-5 with higher scores indicating greater follow-up/coordination).
Combined items from the Treatment Burden Questionnaire (TBQ) that appear to measure similar constructs. | 6-12 Months
  Items that assess self-management tasks (3 items that range from 0-30 with lower scores indicating less self-management burden), medical visits (2 items that range from 0-20 with lower scores indicating less burden from doctor visits), laboratory tests and other examinations (1 item that ranges from 0-10 with lower scores indicating less burden from lab exams), relationships with providers (1 item with scores ranging from 0-10 with lower scores indicating less burden from relationships with providers), medications (4 items with scores ranging from 0-40 with lower scores indicating less burden from medications).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tinetti ME, Naik AD, Dindo L, Costello DM, Esterson J, Geda M, Rosen J, Hernandez-Bigos K, Smith CD, Ouellet GM, Kang G, Lee Y, Blaum C. Association of Patient Priorities-Aligned Decision-Making With Patient Outcomes and Ambulatory Health Care Burden Among Older Adults With Multiple Chronic Conditions: A Nonrandomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1688-1697. doi: 10.1001/jamainternmed.2019.4235. PMID 31589281

DOCUMENTS (1):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03600389/Prot_000.pdf